CLINICAL TRIAL: NCT07160439
Title: Evaluating Digital Micro-Interventions to Reduce Distress and Increase Wellbeing in Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Philip Chow, Ph.D., Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6002; 4R37CA248434-05 (NIH)
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Mental Health Issue; Breast Cancer
Keywords: Depression; Anxiety; Well-Being
MeSH Terms: conditions — Breast Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Pilot study to test early stage digital micro-interventions (n=20 per micro-intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Savoring (Experimental): Participants are asked to think of a positive and personally meaningful memory to meditate on. They are led through steps to enter their memory, which is then summarized and turned into a meditation practice.
  Interventions: Behavioral: Digital Micro-Interventions
- Gratitude (Experimental): Participants are asked to generate a list of things they are grateful for. They are led through an automated process of selecting a source of gratitude and reflecting on it.
  Interventions: Behavioral: Digital Micro-Interventions
- Challenging UnhelpfulThoughts (Experimental): Participants are taught how to identify unhelpful thoughts, challenge them, and generate more balanced, helpful thoughts through an automated process that leads them step-by-step.
  Interventions: Behavioral: Digital Micro-Interventions
- Psychoeducation (Experimental): Participants receive access to psychoeducation content on mental health, distress, and well-being. They are provided tidbits of information every day to learn from.
  Interventions: Behavioral: Digital Micro-Interventions
- Behavioral Activation (Experimental): Participants are led through an automated process of identifying tasks they can accomplish in their daily lives.
  Interventions: Behavioral: Digital Micro-Interventions
- Acceptance (Experimental): Participants are led through an automated process of accepting, rather than actively trying to push away, their distressing emotions or thoughts.
  Interventions: Behavioral: Digital Micro-Interventions

INTERVENTIONS:
Behavioral: Digital Micro-Interventions — Digital Micro-Interventions are brief interventions that target specific behavioral and cognitive mechanisms of mental health, designed for brief periods of engagement.

SUMMARY:
Digital mental and behavioral health interventions have potential to significantly improve accessibility for the large number of breast cancer survivors who need treatments. However, the landscape of digital interventions tested in this population remains limited, with the few that have been tested primarily focused on reducing symptoms of mental disorders. This is problematic given the range of psychosocial needs among breast cancer survivors, including those who may not have active mental health symptoms, yet could benefit from learning effective coping skills. Moreover, all of these interventions follow a "one size fits all" approach, lacking precision in terms of when, where, and to whom they should be given. The overarching goals of this project are to develop and pilot a variety of digital micro-interventions (DMIs) for breast cancer survivors - highly focused, technology-enabled interventions that can be delivered in the context of a person's daily life with little burden on the individual.

ELIGIBILITY:
Inclusion Criteria:

* Age = 18 years.
* 0-5 years post-diagnosis of Stage I, II, or III female breast cancer.
* Elevated symptoms of depression and/or anxiety as measured by the PHQ-8 (score > 9) or GAD-7 (score > 7).

Exclusion Criteria:

* Receiving individual (1 on 1) treatment for depression and/or anxiety to avoid treatment interference (note, individuals will be permitted to enroll if they are taking antidepressant medication and have not had an appointment to adjust the dosage over the past 2 weeks)
* Active suicidal ideation during the enrollment/screening call based on a trained staff member orally administering the suicidality item from the PHQ-9 to individuals on the phone ("In the last 2 weeks, have you had thoughts that you would be better off dead, or thoughts of hurting yourself in some way?"). If an individual responds in any way other than "not at all" based on the available response options (i.e., either "several days", "more than half the days", or "nearly every day"), or if they mention having suicidal ideation or thoughts of death during the enrollment/screening call, the Pitt-Optimum risk assessment tool will be administered. Only participants deemed low risk may proceed in enrollment; all will be given additional resources.
* Do not have an app-compatible phone (i.e., iOS 10.3 or later or Android 4.0.3 or later).
* Cannot read and speak English (interventions only available in English).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Digital Micro-Intervention | Post 1 week
  12 item scale measuring satisfaction and acceptability. Each question is scored on a 0-4 scale with a total raw summed score range of 0-48. Higher scores indicate greater satisfaction and acceptability.

SECONDARY OUTCOMES:
PROMIS-29 Profile | Baseline
  28 items that measure aspects of physical and mental health. Each question is scored on a 1-5 scale with a total raw score range of 28-140. Higher scores indicate worse overall health. A 29th item that assesses pain from 1-10 was omitted to limit redundancy with another pain measure.
PROMIS-29 Profile | Post 1 week
  28 items that measure aspects of physical and mental health. Each question is scored on a 1-5 scale with a total raw score range of 28-140. Higher scores indicate worse overall health. A 29th item that assesses pain from 1-10 was omitted to limit redundancy with another pain measure.
Pain, Enjoyment of Life and General Activity (PEG) Scale | Baseline
  Assesses chronic pain based on 3 items, each one ranging from 0-10. Scores range from 0-30, with higher scores indicating more pain severity and interference.
Pain, Enjoyment of Life and General Activity (PEG) Scale | Post 1 week
  Assesses chronic pain based on 3 items, each one ranging from 0-10. Scores range from 0-30, with higher scores indicating more pain severity and interference.
Emotion Regulation Questionnaire | Baseline
  A 10 item scale to reassess for two emotion regulation strategies: cognitive reappraisal and expressive suppression. Participants rate each item on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree). Scores for each subscale range from 1-7 (after dividing by the number of items), with higher scores indicating a greater tendency to use that particular emotion regulation strategy.
Emotion Regulation Questionnaire | Post 1 week
  A 10 item scale to reassess for two emotion regulation strategies: cognitive reappraisal and expressive suppression. Participants rate each item on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree). Scores for each subscale range from 1-7 (after dividing by the number of items), with higher scores indicating a greater tendency to use that particular emotion regulation strategy.
Insomnia Severity Index | Baseline
  A 7-item measure to evaluate severity of insomnia symptoms. Each item is evaluated on a scale from 0-4. Scores range from 0-28, with higher scores indicating greater severity of insomnia symptoms.
Insomnia Severity Index | Post 1 week
  A 7-item measure to evaluate severity of insomnia symptoms. Each item is evaluated on a scale from 0-4. Scores range from 0-28, with higher scores indicating greater severity of insomnia symptoms.
Patient Health Questionnaire-8 | Baseline
  8 item scale that measures depression symptoms on a continuous scale. Scores range from 0-24, with a higher score indicating greater severity of symptoms of depression.
Patient Health Questionnaire-8 | Post 1 week
  8 item scale that measures depression symptoms on a continuous scale. Scores range from 0-24, with a higher score indicating greater severity of symptoms of depression.
Generalized Anxiety Disorder-7 | Baseline
  7 item scale that measures anxiety symptoms on a continuous scale. Scores range from 0-21, with a higher score indicating greater severity of symptoms of anxiety.
Generalized Anxiety Disorder-7 | Post 1 week
  7 item scale that measures anxiety symptoms on a continuous scale. Scores range from 0-21, with a higher score indicating greater severity of symptoms of anxiety.

OTHER OUTCOMES:
Qualitative Interview | Post 1 week
  Remote interview to assess for participant feedback on usability, obstacles to use, and suggestions for improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No